CLINICAL TRIAL: NCT06240910
Title: Effects of Aerobic Training and Neurodynamics to Prevent Fall and Improve Balance in Patients With Diabetic Neuropathy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/23/0236
Record Dates: First submitted 2024-01-28; First posted 2024-02-05 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2024-01

CONDITIONS: Diabetic Neuropathies
Keywords: Aerobic exercise training; Balance and fall; Diabetic neuropathy; Neural mobilization
MeSH Terms: conditions — Diabetic Neuropathies

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neurodynamics (Experimental): Neuro dynamics involving Stretching and gliding of the Sciatic nerve (performing each exercise for 30 s at a slow and comfortable pace of 1 repetition per ~3-4 s. The participants rested for 60 s between each exercise. The total duration of the interventions was approximately 10 min.).The whole treatment session on a single day will be of 40-60 minutes of duration (involving both aerobic exercise + neurodynamics) 3. times a week for 6 weeks according to the American diabetes association, accumulating a minimum of 150 minutes/week.
  Interventions: Other: Neurodynamics
- Aerobic training (Experimental): Aerobic exercise will involve warm-up by stretching and flexibility exercises for 5 minutes, Treadmill walking for 6 minutes, and Stationary bicycle for 6 minutes
  Interventions: Other: Aerobic training

INTERVENTIONS:
Other: Neurodynamics — Neuro dynamics involving Stretching and gliding of the Sciatic nerve (performing each exercise for 30 s at a slow and comfortable pace of 1 repetition per ~3-4 s. The participants rested for 60 s between each exercise.
  Arms: Neurodynamics
Other: Aerobic training — Aerobic exercise will involve warm-up by stretching and flexibility exercises for 5 minutes, Treadmill walking for 6 minutes, and Stationary bicycle for 6 minutes
  Arms: Aerobic training

SUMMARY:
Diabetes is a group of metabolic diseases, characterized by hyperglycemia resulting from defects in insulin secretion, actionor both. The chronic hyperglycemia of diabetes is associated with long-term damage, dysfunction, and failure of differentorgans, especially the eyes, kidneys, nerves, heart, and blood vessels. In long standing cases of both diabetes type 1 and 2, about 60 % individuals had diabetic neuropathy. Patients suffering from diabetes are more prone to fall, possibly due to balance issues and sensory ataxia.

DETAILED DESCRIPTION:
This study will be a Randomized controlled trial. Participants who have DM2 for past 7 years and who score >2/13 on Michigan neuropathy screening instrument questionnaire with at least 2 DPN symptoms will be screened for this study. Participants with any fracture in lower limb , complete loss of foot perception, comorbidities, using assistive devices and already involved in structured physiotherapy interventional program will be excluded from this randomized controlled trial study. Participants will be selected with non-probability consecutive sampling and will be randomly allocated using computer generated randomizer in two groups i.e., experimental group and control group. Balance and risk of fall will be assessed through Berg Balance scale, functional reach test , Romberg test and morse fall scale before and after giving interventions. Treatment session will be given 3 days a week for 6 weeks. Participants in control group will be given neurodynamics for sciatic nerve ( the total duration of interventions will be approximately 10 minutes a day for 3 days in a week for 6 weeks. Experimental group will be given aerobic exercise interventions (involving warm-up by stretching and flexibility exercisesfor 5 minutes, treadmill walking and stationary bicycle training with 6 minutes a day for 3 days in a week for 6 weeks) along with neural mobilization for sciatic nerve ( 10 minutes a day for 3 days in a week for 6 weeks), so the total duration of interventions for experimental group will be 40-60 minutes a day for 3 days in a week for 6 weeks. Given the high prevalence and substantial impact of diabetic neuropathy on balance and fall risk, it is imperative to explore effective interventions (aerobic exercise + neurodynamics) for managing these impairments. Individuals may experience improved proprioception, enhanced muscle coordination, and optimized neural tissue mobility, leading to reduced fall risk and improved functional independence. Data will be analyze using SPSS 23.

ELIGIBILITY:
Inclusion Criteria:

Age ranged between 45-67 years.

* Both male and female genders
* DM for the past 7 years.
* Scored >2/13 on Michigan neuropathy screening instrument (MNSI) questionnaire including at least two DPN symptoms.

Exclusion Criteria:

fracture(s) in the lower limb.

* Any participant who suffered from foot ulcers.
* Unstable heart disease, co- Morbid conditions limiting exercise
* inability of subjects to understand and/or co-operate during quantitative sensory testing or manual/nerve mobility testing and/or treatment.
* Any level of physical activity i.e 150 minutes/week
* Receiving any structured supervised physiotherapy interventions.

Ages: 45 Years to 67 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2023-07-17 (Actual); Primary Completion 2024-02-12 (Estimated); Study Completion 2024-02-12 (Estimated)

PRIMARY OUTCOMES:
Berge balance scale | 6 weeks
  The Berg Balance Scale (BBS) is used to objectively determine a patient's ability (or inability) to safely balance during a series of predetermined tasks.

SECONDARY OUTCOMES:
Functional reach test | 6 weeks
  Functional Reach Test (FRT) is a clinical outcome measure and assessment tool for ascertaining dynamic balance in one simple task.

OTHER OUTCOMES:
Morse scale | 6 weeks
  This scale was published by Morse in 1989 and consists of six criteria for assessing the risk of falls: history of falling, secondary diagnosis, ambulatory aid, intravenous therapy/heparin lock, gait, and mental status.
Romberg test | 6 weeks
  The Romberg test is a test that measures a persons sense of balance. Specifically, the test assesses the function of the dorsal column of the spinal cord (the dorsal column is responsible for proprioception).
Michigan neuropathy screening instrument questionnaire | 6 weeks
  The Michigan Neuropathy Screening Instrument (MNSI) is a valid screening tool for DN(19).
  The maximum score of the foot examination is 8 points and a score of equal to or greater than 2 is positive for DPN.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Asrar Yousaf, Principal Investigator — Riphah International University
Locations (2):
- Pakistan (2):
  - Ripha international university, Lahore, Punjab Province
  - Riphah international university, Lahore, Punjab Province

IPD SHARING:
Plan to Share IPD: No